CLINICAL TRIAL: NCT03486756
Title: Internet-delivered Cognitive Behavior Therapy for Asthma-related Anxiety: A Feasibility Study
Brief Title: Internet-delivered CBT for Asthma-related Anxiety: Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Catarina Almqvist Malmros, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MANTRA02
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Asthma
Keywords: Asthma; Anxiety; Stress
MeSH Terms: conditions — Asthma; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is an uncontrolled feasibility study with one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-CBT (Experimental): Internet-CBT for anxiety-related asthma 8 weekly modules of CBT delivered over the internet and targeting enhanced function and decreased symptoms of anxiety. Participants work independently from home with the treatment and receive support from experienced Internet-CBT Psychologists through written messages in the secure platform.
  Interventions: Behavioral: Internet-CBT for anxiety-related asthma

INTERVENTIONS:
Behavioral: Internet-CBT for anxiety-related asthma — The specific assignments in the intervention will be based on individual behavior analysis for each participant.

SUMMARY:
This is a study to investigate acceptability and feasibility of a novel protocol on exposure-based CBT for asthma-related fear delivered over the Internet (Internet-CBT).

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases around the world, with a high prevalence of anxiety disorders. In a prior study (ClinicalTrials.gov ID: NCT03158194) a protocol for exposure-based CBT was developed for asthma-related anxiety. The aim of the current study is to evaluate acceptability and feasibility of our protocol for asthma-related fear when delivered over the Internet (Internet-CBT). The plan is to include 30 participants that will all receive the intervention in this uncontrolled feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* asthma diagnosed by a physician
* anxiety or stress related to asthma

Exclusion Criteria:

* severe psychiatric disorder
* chronic obstructive pulmonary disease (COPD) and other chronic airway disorders other than asthma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Catastrophizing about asthma Scale | Baseline to 8 weeks; baseline to 16 weeks; baseline to 24 weeks.
  Change in catastrophizing cognitions about asthma measured with a self-rating scale at baseline, 8 weeks, 16 weeks and 24 weeks for analysis of effect.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire | Baseline to 8 weeks; baseline to 16 weeks; baseline to 24 weeks.
  Change in subjective worry measured with a self-rating scale measured with a self-rating scale at baseline, 8 weeks, 16 weeks and 24 weeks for analysis of effect.
Asthma control test | Baseline to 8 weeks; baseline to 16 weeks; baseline to 24 weeks.
  Change in asthma control measured with a self-rating scale at baseline, 8 weeks, 16 weeks and 24 weeks for analysis of effect.
Asthma Quality of Life Questionnaire | Baseline to 8 weeks; baseline to 16 weeks; baseline to 24 weeks.
  Change in asthma-related quality of life measured with a self-rating scale at baseline, 8 weeks, 16 weeks and 24 weeks for analysis of effect.
Short Health Anxiety Inventory (SHAI) | Baseline to 8 weeks; baseline to 16 weeks; baseline to 24 weeks.
  Change in health anxiety measured with a self-rating scale at baseline, 8 weeks, 16 weeks and 24 weeks for analysis of effect.
Perceived Stress Scale | Baseline to 8 weeks; baseline to 16 weeks; baseline to 24 weeks.
  Change in perceived stress measured with a self-rating scale at baseline, 8 weeks, 16 weeks and 24 weeks for analysis of effect.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Almqvist Malmros, MD PhD, Principal Investigator — Department of Medical Epidemiology and Biostatistics, Karolinska Institutet
Locations (1):
- Department of Medical Epidemiology and Biostatistics, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonnert M, Sarnholm J, Andersson E, Bergstrom SE, Lalouni M, Lundholm C, Serlachius E, Almqvist C. Targeting excessive avoidance behavior to reduce anxiety related to asthma: A feasibility study of an exposure-based treatment delivered online. Internet Interv. 2021 Jun 17;25:100415. doi: 10.1016/j.invent.2021.100415. eCollection 2021 Sep. PMID 34401374